CLINICAL TRIAL: NCT07192159
Title: Evaluation of a Quantitative Ultrasound Model(DeepUSFF) for Liver Fat Quantification in Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease: A Multicenter Prospective Study Using MRI-PDFF as the Reference Standard
Brief Title: Quantitative Ultrasound(DeepUSFF) vs MRI-PDFF for Liver Fat Assessment in MASLD
Acronym: DeepUSFF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Northeastern Ohio Radiology Research and Education Fund (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2503-162-1625
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Hepatic Steatosis; Liver Disease Parenchymal
Keywords: Metabolic dysfunction-associated steatotic liver disease; Quantitative ultrasound; MRI-PDFF; Liver fat quantification; Hepatic steatosis; Deep learning
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Intervention Model Description: Single Group Cross-Sectional Diagnostic Accuracy Study All enrolled participants will undergo both diagnostic procedures (quantitative ultrasound and MRI-PDFF) within a 7-day window to minimize temporal variation in liver fat content. This single-group design allows for direct paired comparison between the two diagnostic methods in the same participants, eliminating inter-subject variability and providing optimal conditions for correlation analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Quantitative Ultrasound Fat Fraction Assessment (Experimental): All enrolled participants undergo two non-invasive diagnostic imaging procedures within a 7-day window for direct comparison of liver fat quantification methods:
  1. **Quantitative Ultrasound Examination**: Performed using Samsung RS85 ultrasound system with CA1-7S convex probe to obtain ultrasound fat fraction (DeepUSFF). The examination includes standard liver ultrasound assessment followed by quantitative fat fraction measurements in the right hepatic lobe (S5 or S8 segments). Multiple measurements (5 per session) are obtained during breath-holding to ensure reproducibility. Total examination time: approximately 10-15 minutes.
  2. **Non-contrast Liver MRI with PDFF**: Magnetic resonance imaging with proton density fat fraction (MRI-PDFF) sequence and MR elastography performed within 7 days of the ultrasound examination. The MRI protocol includes breath-hold sequences (10-20 seconds each) for optimal image quality. Total examination time: approximately 15 minutes.
  Interventions: Device: Quantitative ultrasound (DeepUSFF)

INTERVENTIONS:
Device: Quantitative ultrasound (DeepUSFF) — **Novel Quantitative Ultrasound Technology Assessment**
  This study evaluates Samsung Medison's proprietary DeepUSFF (Deep Learning-based Ultrasound Fat Fraction) technology, a next-generation quantitative ultrasound method for liver fat assessment that differs from conventional ultrasound approaches in several key aspects: advanced RF data analysis, proprietary technology, standardized protocol, direct MRI-PDFF correlation, specific MSALD poopulation and multicenter design.

SUMMARY:
This multicenter prospective study aims to evaluate the correlation between quantitative ultrasound fat fraction (USFF) and MRI-PDFF (Proton Density Fat Fraction) for liver fat quantification in patients with metabolic dysfunction-associated steatotic liver disease (MASLD). The study will compare the diagnostic accuracy of quantitative ultrasound imaging against MRI-PDFF as the reference standard.

DETAILED DESCRIPTION:
Background: Metabolic dysfunction-associated steatotic liver disease (MASLD) is a common liver disease requiring accurate assessment for treatment planning and monitoring. While liver biopsy remains the gold standard, it is invasive with potential complications. MRI-PDFF has emerged as an accurate non-invasive method, but it is expensive and has limited accessibility. Quantitative ultrasound techniques using RF data have been developed to provide objective liver fat assessment.

Objective: To prospectively evaluate the correlation between quantitative ultrasound-derived fat fraction (DeepUSFF) and MRI-PDFF in patients with suspected MASLD across different ethnicities and varying degrees of hepatic steatosis.

Methods: This prospective multicenter study will recruit 62 patients (31 from each participating center) suspected of having MASLD. All participants will undergo both quantitative ultrasound examination and non-contrast liver MRI within one week. The primary endpoint is the correlation coefficient between ultrasound fat fraction and MRI-PDFF. Secondary endpoints include diagnostic accuracy metrics and inter-observer reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected MASLD based on abnormal ultrasound or liver function tests requiring liver ultrasound or MRI examination
* BMI ≥25 kg/m² or waist circumference >90 cm (male) or >80 cm (female), suggesting high likelihood of fatty liver disease
* Living liver transplant donors requiring preoperative liver ultrasound or MRI examination
* Age ≥18 years
* Understanding and signing informed consent

Exclusion Criteria:

* Significant alcohol consumption in the past 2 years:

Male: ≥30-60g/day average alcohol intake Female: ≥20-50g/day average alcohol intake

-Chronic liver disease:

Histological diagnosis of chronic liver disease HBsAg positive Anti-HCV positive Other suspected chronic liver diseases

-Liver failure:

Serum albumin <3.2 g/dL INR >1.3 Direct bilirubin >1.3 mg/dL

* History of esophageal varices, ascites, hepatic encephalopathy, or acute biliary obstruction
* History of liver cancer diagnosis or treatment
* History of liver surgery
* Pregnancy
* Inability to obtain adequate liver ultrasound imaging:

Patient cooperation impossible Inadequate image acquisition as determined by investigator

-Inability to obtain adequate liver MRI imaging: Patient cooperation impossible Severe obesity preventing MRI examination MRI contraindications (cardiac pacemaker, etc.) Other factors preventing adequate imaging as determined by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between Ultrasound Fat Fraction and MRI-PDFF | At enrollment (single time point assessment)
  earson correlation coefficient between quantitative ultrasound fat fraction (USFF) and MRI-PDFF
Correlation between Ultrasound Fat Fraction and MRI-PDFF | At enrollment (single time point assessment)
  Measure: Pearson correlation coefficient between quantitative ultrasound fat fraction (USFF) and MRI-PDFF

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital; Richard Gary Barr, MD, Study Director — Northeastern Ohio Radiology Research and Education Fund
Locations (2):
- southwoods imaging (Northeastern Ohio Radiology Research and Education Fund ), Boardman, Ohio, United States
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified quantitative ultrasound measurements (USFF values) De-identified MRI-PDFF measurements Anonymized clinical variables (age, BMI, laboratory values) Statistical analysis datasets without patient identifiers
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months following article publication
Access Criteria: Requests should be directed to the corresponding author with a detailed research proposal Data sharing agreements will be required Institutional review board approval may be required for secondary analyses
URL: https://snuh.org/research/data-sharing-policy

REFERENCES:
- [Background] Xie WJ, Zhang B. Learning the Formation Mechanism of Domain-Level Chromatin States with Epigenomics Data. Biophys J. 2019 May 21;116(10):2047-2056. doi: 10.1016/j.bpj.2019.04.006. Epub 2019 Apr 11. PMID 31053260
- [Background] Fan C, Shen M, Nussinov Z, Liu Z, Sun Y, Liu YY. Reply to: Deep reinforced learning heuristic tested on spin-glass ground states: The larger picture. Nat Commun. 2023 Sep 14;14(1):5659. doi: 10.1038/s41467-023-41108-w. No abstract available. PMID 37709759
- [Background] Zhou G, Qin Y, Petticord D, Qiao X, Jiang M. Plant-ant interactions mediate herbivore-induced conspecific negative density dependence in a subtropical forest. Sci Total Environ. 2024 Jun 1;927:172163. doi: 10.1016/j.scitotenv.2024.172163. Epub 2024 Apr 1. PMID 38569958